CLINICAL TRIAL: NCT05377879
Title: A Clinical Trial to Determine the Effectiveness of Using the Proposed Decision Support Tool for Each Patient's Customized Optimal Drug Dosage Profile
Brief Title: An Advanced Decision Support Tool for Personalized Medicine for IVF Using Modeling and Optimization
Acronym: OPT-IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stochastic Research Technologies LLC (Industry)
Collaborators: Akansha Hospital and Research Institute, India (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: opivf-protocol-22-1
Record Dates: First submitted 2022-05-04; First posted 2022-05-17 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: IVF

STUDY DESIGN:
Intervention Model Description: OPT-IVF is a decision support tool which personalizes and optimizes dosage for each patient for each cycle.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Identity of the patient in any form is not provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPTIVF predicted drug dosage (Experimental): In our study, we will be using the patient's age and day three serum day AMH and FSH levels to decide the starting dose for the patient's cycle. We will use the first two days of data collected (Follicular size distribution, estrogen levels) for that patient to determine the optimal dosage profile for the entire cycle for that patient with the help of the decision support tool OPTIVF for this intervention in the clinical trial.
  Interventions: Device: OPT-IVF dosage
- Traditional drug treatment (No Intervention): Patients where drug dosage is decided by the physician based on ultrasound and estrogen levels for each day of the cycle.

INTERVENTIONS:
Device: OPT-IVF dosage — Dosage predicted for each patient by the decision support tool OPTIVF
  Arms: OPTIVF predicted drug dosage

SUMMARY:
Aim: A Clinical trial to determine the effectiveness of using the proposed decision support tool (OPTIVF) for each patient's customized optimal drug dosage profile. This will be a two-arm (in the ratio 1:3) clinical trial involving more than 80 participants; one arm will undergo superovulation using dosages predicted by the decision support tool while the other arm has undergone current standard treatment. The investigators will compare the outcomes of the two groups of participants in terms of the numbers and percentage of mature follicles retrieved at the end of each cycle, total FSH and HMG dosages used, and the number of required testing days for that cycle. The participants considered will include all ages, with and without PCOS, and low, average, and high responders.

DETAILED DESCRIPTION:
This is a multi-site cohort with two arms (one arm for the intervention and one arm for the traditional approach) clinical trial involving more than 70 participants. The population size for the clinical trial was kept small because retrospective data for 170 patients is already collected each for comparing the two arms of the trial. Further, the data for 45 patients is there from the early small clinical trial we conducted in India.

The main site for this task is the Akansha Hospital, India, and all the analysis will be carried out at the Stochastic Research site. Dr. Urmila Diwekar will be an investigator from the Stochastic Research Technologies LLC, and Dr. Nayana Patel will be an investigator from Akansha Hospital and Research Institute.

In our study, the investigators will be using the participant's age and day three serum day AMH and FSH levels to decide the starting dose for the patient's cycle. The investigators will use the first two days of data collected (Follicular size distribution, estrogen levels) for that paticipant to determine the optimal dosage profile for the entire cycle for that participant with the help of the decision support tool OPT-IVF for this intervention in the clinical trial.

Primary and secondary outcomes will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing infertility treatment

Exclusion Criteria:

* No male participants

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a treatment for women only
Enrollment: 44 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of follicles retrieved | At the end of cycle 1 (each cycle ranges from 10 to 12 days)
  follicles retrieved
Number of M2s | At the end of cycle 1(each cycle ranges from 10 to 12 days)
  Number of M2s retrieved
No. of Very Good Embryos | At the end of cycle 1 (each cycle ranges from 10 to 12 days)
  Grade A Embryos

SECONDARY OUTCOMES:
Pregnancy | 9 to 12 days after the transfer
  Whether pregnancy is resulted or not

CONTACTS AND LOCATIONS:
Overall Officials: Urmila Diwekar, Ph.D., Principal Investigator — Stochastic Research Technologies/University of Illinois at Chicago
Locations (1):
- Akansha Hospital and Research Institute, Anand, Gujarat, India

IPD SHARING:
Plan to Share IPD: Yes
Please contact urmila@vri-custom.org for IPD.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Available now.
Access Criteria: Please contact urmila@vri-custom.org for IPD.

REFERENCES:
- [Background] Nisal A, Diwekar U, Bhalerao V. Personalized medicine for in vitro fertilization procedure using modeling and optimal control. J Theor Biol. 2020 Feb 21;487:110105. doi: 10.1016/j.jtbi.2019.110105. Epub 2019 Dec 3. PMID 31809718
- [Background] Yenkie KM, Diwekar UM, Bhalerao V. Modeling the superovulation stage in in vitro fertilization. IEEE Trans Biomed Eng. 2013 Nov;60(11):3003-8. doi: 10.1109/TBME.2012.2227742. Epub 2012 Nov 15. PMID 23193444
- [Background] Yenkie KM, Diwekar U. Uncertainty in clinical data and stochastic model for in vitro fertilization. J Theor Biol. 2015 Feb 21;367:76-85. doi: 10.1016/j.jtbi.2014.11.004. Epub 2014 Dec 4. PMID 25484007
- See also: description is available at http://www.stochastic-research.com/InVitroFertilization.html — http://www.stochastic-research.com